CLINICAL TRIAL: NCT00829725
Title: Randomized, Prospective, Multi-center, Comparison Study of 3-4-screws-internal Fixation With Multi-screw-system Targon FN for Femoral Neck Fracture
Brief Title: Comparison Study of 3-4-screws-internal Fixation With Multi-screw-system Targon FN for Femoral Neck Fracture
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Nahshon Shazar MD. Head Trauma Unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-5569-NS-CTIL
Record Dates: First submitted 2009-01-25; First posted 2009-01-27 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Femoral Neck Fractures
Keywords: subcapital femoral fractures; transcervical femoral fractures; TARGON FN
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- screws-internal fixation (Active Comparator): 3-4-screws-internal fixation
  Interventions: Device: screws-internal fixation
- TARGON FN (Experimental): The Targon FN implant consists of a small side plate with six locking screw ports. The two distal holes are used to fix the plate to the lateral cortex of the femur with angle stable 4.5 mm cortical screws. The proximal holes allow the implementation of up to four "TeleScrews" which cross the fracture site. These 6.5 mm screws are dynamic and allow therewith the collapse of the fracture at the femoral neck. The sliding during the collapse occurs within these screws so that a protrusion of the screws in the lateral soft tissue is prevented
  Interventions: Device: TARGON FN

INTERVENTIONS:
Device: screws-internal fixation — 3-4-screws-internal fixation
  Arms: screws-internal fixation
Device: TARGON FN — The Targon FN implant consists of a small side plate with six locking screw ports. The two distal holes are used to fix the plate to the lateral cortex of the femur with angle stable 4.5 mm cortical screws. The proximal holes allow the implementation of up to four "TeleScrews" which cross the fracture site. These 6.5 mm screws are dynamic and allow therewith the collapse of the fracture at the femoral neck. The sliding during the collapse occurs within these screws so that a protrusion of the screws in the lateral soft tissue is prevented
  Arms: TARGON FN

SUMMARY:
The purpose of this study is to compare between two methods of internal fixation, the 3-4 parallel screws or the Targon FN implant in gardens type 1-2 or Pauwels type 1-2 femoral neck fractures in terms of the outcomes and complications associated with the treatment of these fractures.

DETAILED DESCRIPTION:
Intracapsular femoral neck fractures include subcapital and transcervical fractures. They typically occur in a bimodal age distribution, with most occurring in the elderly population. The rest are the result of high energy injury in the young. Undisplaced hip fractures are defined as fractures where the inferior cortical buttress is undisplaced on the anteroposterior (AP) radiograph.[1] Undisplaced hip fractures includes fractures impacted in all degrees of valgus regardless of any angulations at the fractures' edges seen on the lateral radiographs. The fractures can be classified using either the Garden or Pauwel classifications for subcapital fracture or transcervical fractures, respectively. The choice of treatment of undisplaced hip fractures is contentious, especially in elderly patients. The options range from nonoperative treatment in younger patients with stable impacted fractures to primary hemiarthroplasty for frail, elderly patients.[2] Although some of those fracture, like impacted valgus fractures have a degree of inherent stability, internal fixation is generally recommended because nonunion rates of up to 39% have been reported with nonsurgical treatment. [3] In one study the authors examined 375 patients with nondisplaced intracapsular fractures treated with internal fixation [cannulated cancellous screws (366 patients), dynamic hip screws (nine patients)]. The authors noted a nonunion rate of 6.4% and an osteonecrosis rate of 4.0%. Age, walking ability, degree of impaction evident on the anteroposterior radiograph, and angulation on the lateral radiograph were determined to be predictive of healing complications. In this study, the conversion rate to arthroplasty was 7.7%. [4] Femoral neck fractures in young adults are associated with higher incidences of femoral head osteonecrosis [5-13] and nonunion [5, 6, 9, 14]. The reported rate of osteonecrosis after a femoral neck fracture in young patients ranges from 12% to 86% [5, 8-17]. This complication may lead to collapse of the femoral head and osteoarthritis. Salvage procedures, such as osteotomy, and other reoperations have high failure rates, and arthroplasty procedures are not ideal, given the patient's young age and higher level of activity. The achievement of an anatomic reduction and stable internal fixation is imperative. The Targon FN implant consists of a small side plate with six locking screw ports. The two distal holes are used to fix the plate to the lateral cortex of the femur with angle stable 4.5 mm cortical screws. The proximal holes allow the implementation of up to four "TeleScrews" which cross the fracture site. These 6.5 mm screws are dynamic and allow therewith the collapse of the fracture at the femoral neck. The sliding during the collapse occurs within these screws so that a protrusion of the screws in the lateral soft tissue is prevented.

The only report was reported by Martyn Parker MD and was released in Jatros Orthopädie 2008. He reported a serial of 50 femoral neck fractures, 27 (54%) of the fractures were undisplaced and 23 (48%) were displaced. There were two cases of fracture non-union, In one patient the plate became detached. One patient with a non-displaced femur neck fracture showed early radiographic signs of a possible avascular necrosis after one year. The implant was removed and the symptoms improved somewhat.

The purpose of this study is therefore to compare between two methods of internal fixation, the 3-4 parallel screws or the Targon FN implant in gardens type 1-2 or Pauwels type 1-2 femoral neck fractures in terms of the outcomes and complications associated with the treatment of these fractures. we expect around 5% complications using the Targon FN implant comparing to 11% complications with the screws.

ELIGIBILITY:
Inclusion Criteria:

* nondisplaced subcapital femoral fracture (gARDEN 1-2)
* transcervical femoral fractures(Pauwells 1 & 2).
* Fractures operated within 7 days
* ASA score 1-3

Exclusion Criteria:

* prior hip surgery
* pathological fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
overall survival, fixation survival and a composite end-point combining the two | 1 year

SECONDARY OUTCOMES:
length of surgery, bleeding, ambulation | 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Meir Medical Center, Kfar Saba
  - Sheba medical center, Tel Litwinsky
  - Assaf-Harofeh Medical Center, Zrifin

REFERENCES:
- [Background] Hui AC, Anderson GH, Choudhry R, Boyle J, Gregg PJ. Internal fixation or hemiarthroplasty for undisplaced fractures of the femoral neck in octogenarians. J Bone Joint Surg Br. 1994 Nov;76(6):891-4. PMID 7983113
- [Background] Tanaka J, Seki N, Tokimura F, Hayashi Y. Conservative treatment of Garden stage I femoral neck fracture in elderly patients. Arch Orthop Trauma Surg. 2002 Feb;122(1):24-8. doi: 10.1007/s004020100318. PMID 11995876
- [Background] Conn KS, Parker MJ. Undisplaced intracapsular hip fractures: results of internal fixation in 375 patients. Clin Orthop Relat Res. 2004 Apr;(421):249-54. PMID 15123955
- [Background] Protzman RR, Burkhalter WE. Femoral-neck fractures in young adults. J Bone Joint Surg Am. 1976 Jul;58(5):689-95. PMID 932067
- [Background] Dedrick DK, Mackenzie JR, Burney RE. Complications of femoral neck fracture in young adults. J Trauma. 1986 Oct;26(10):932-7. doi: 10.1097/00005373-198610000-00013. PMID 3773004
- [Background] Zetterberg CH, Irstam L, Andersson GB. Femoral neck fractures in young adults. Acta Orthop Scand. 1982 Jun;53(3):427-35. doi: 10.3109/17453678208992237. PMID 7090765
- [Background] Swiontkowski MF, Winquist RA, Hansen ST Jr. Fractures of the femoral neck in patients between the ages of twelve and forty-nine years. J Bone Joint Surg Am. 1984 Jul;66(6):837-46. doi: 10.2106/00004623-198466060-00003. PMID 6736085
- [Background] Kofoed H. Femoral neck fractures in young adults. Injury. 1982 Sep;14(2):146-50. doi: 10.1016/0020-1383(82)90049-3. PMID 7141676
- [Background] Shih CH, Wang KC. Femoral neck fractures. 121 cases treated by Knowles pinning. Clin Orthop Relat Res. 1991 Oct;(271):195-200. PMID 1914295
- [Background] Lee CH, Huang GS, Chao KH, Jean JL, Wu SS. Surgical treatment of displaced stress fractures of the femoral neck in military recruits: a report of 42 cases. Arch Orthop Trauma Surg. 2003 Dec;123(10):527-33. doi: 10.1007/s00402-003-0579-8. Epub 2003 Sep 2. PMID 12955538
- [Background] Visuri T, Vara A, Meurman KO. Displaced stress fractures of the femoral neck in young male adults: a report of twelve operative cases. J Trauma. 1988 Nov;28(11):1562-9. doi: 10.1097/00005373-198811000-00007. PMID 3184218
- [Background] Haidukewych GJ, Rothwell WS, Jacofsky DJ, Torchia ME, Berry DJ. Operative treatment of femoral neck fractures in patients between the ages of fifteen and fifty years. J Bone Joint Surg Am. 2004 Aug;86(8):1711-6. doi: 10.2106/00004623-200408000-00015. PMID 15292419
- [Background] Upadhyay A, Jain P, Mishra P, Maini L, Gautum VK, Dhaon BK. Delayed internal fixation of fractures of the neck of the femur in young adults. A prospective, randomised study comparing closed and open reduction. J Bone Joint Surg Br. 2004 Sep;86(7):1035-40. doi: 10.1302/0301-620x.86b7.15047. PMID 15446534
- [Background] Tooke SM, Favero KJ. Femoral neck fractures in skeletally mature patients, fifty years old or less. J Bone Joint Surg Am. 1985 Oct;67(8):1255-60. PMID 4055851
- [Background] Gautam VK, Anand S, Dhaon BK. Management of displaced femoral neck fractures in young adults (a group at risk). Injury. 1998 Apr;29(3):215-8. doi: 10.1016/s0020-1383(97)00184-8. PMID 9709424
- [Background] Askin SR, Bryan RS. Femoral neck fractures in young adults. Clin Orthop Relat Res. 1976 Jan-Feb;(114):259-64. PMID 1261119
- [Background] LOW-ANGLE FIXATION IN FRACTURES OF THE FEMORAL NECK R. S. Garden J Bone Joint Surg Br 1961 43-B: 647-663